CLINICAL TRIAL: NCT01320111
Title: Randomised Phase II Study of Paclitaxel Alone Versus Paclitaxel Plus Sorafenib in Second- or Third-line Treatment of Patients With Metastatic Breast Cancer
Brief Title: Breast Cancer Study: Paclitaxel Versus Paclitaxel Plus Sorafenib in Second- or Third-line Treatment
Acronym: PASO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gesellschaft fur Medizinische Innovation - Hamatologie und Onkologie mbH (Other)
Collaborators: iOMEDICO AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GMIHO-008/2008; 2009-018025-73 (EudraCT Number)
Record Dates: First submitted 2011-03-17; First posted 2011-03-22 (Estimated); Last update posted 2017-02-20 (Actual); Status verified 2014-07

CONDITIONS: Metastatic Breast Cancer
Keywords: progression free survival; paclitaxel; sorafenib; metastatic breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Paclitaxel; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1: PA (Active Comparator): patient is treated with paclitaxel only
  Interventions: Drug: Paclitaxel
- Arm 2: PASO (Experimental): patient is treated with paclitaxel AND sorafenib
  Interventions: Drug: Paclitaxel and Sorafenib

INTERVENTIONS:
Drug: Paclitaxel and Sorafenib — intravenous solution, 80 mg/sqm, 3 times per cycle, with one cycle = 28 d and application at days 1, 8 and 15
  AND
  pills (200mg), cycle 1: 400 mg / day cycle 2: 600 mg / day from cycle 3: 800 mg / day
  Other Names: sorafenib = nexavar
  Arms: Arm 2: PASO
Drug: Paclitaxel — intravenous solution, 80 mg/sqm, 3 times per cycle, with one cycle = 28 d and application at days 1, 8 and 15
  Arms: Arm 1: PA

SUMMARY:
AIM OF STUDY

Primary Efficacy Variable:

The primary study objective is the proof of efficacy, measured by progression free survival (PFS) in the treatment of metastatic or locally inoperable recurrent breast cancer.

Progression-free survival (PFS) is defined as the time from randomisation to disease progression or death.

Secondary Efficacy Variables:

* Clinical benefit (CR+PR+SD)
* ORR (CR+PR)
* Time to progression
* Time to next Treatment (TTT)
* Overall survival
* Safety profile

DETAILED DESCRIPTION:
Today breast carcinoma is the leading cancer type and the second frequent cause of cancer death in adult women. This tumor remains a challenge in modern oncology despite recent advances by introducing new classes of chemotherapy like taxanes and antibodies for the HER-2/neu positive tumors. Recently it was shown that the combination of conventional chemotherapy with a monoclonal antibody against VEGF can further increase the response and progression free survival by combination with an antiangiogenic therapy. It is supposed that this effect might result in a prolonged survival.

Sorafenib, a new developed oral inhibitor for tyrosine kinases which are responsible for the signal transduction after binding to the VEGF receptor and the RAS-Raf-MEK-ERK pathway seems efficient in the treatment of a broad range of tumors.

The multi-kinase inhibitor Sorafenib targets the Raf/MEK/ERK pathway at the level of Raf kinase and the receptor tyrosine kinases VEGFR-2 and PDGFR-β, thereby affecting both, the tumour and the vasculature. Preclinical studies as well as phase I trials showed anti-tumour activity in patients with metastatic breast cancer treated with single-agent sorafenib.

This multicentre, phase II, open-label, randomised study is designed to assess the potential prolongation in progression free survival in patients with metastatic breast cancer in combination with standard chemotherapy paclitaxel compared with the paclitaxel monotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed adenocarcinoma of the breast
2. HER-2/neu negative (primary tumour site HER-2/neu negative by ICH/FISH test)
3. Second till third-line of chemotherapy
4. Female, age ≥ 18 years.
5. ECOG Performance Status of 0 or 1 (Karnofsky-Index ≥ 70%)
6. Life expectancy of at least 12 weeks.
7. Subjects with at least one uni-dimensional (for RECIST 1.1) measurable lesion. Lesions must be measured by Xray (pulmonary lesions only) or CT-scan or MRI (Patients with only measurable bone lesions can be also included, as long they meet the criteria for RECIST 1.1.; means, lytic bone lesions or mixed lytic-blastic bone lesions with identifiable soft tissue components.)
8. No prior therapy for locally recurrent or metastatic disease with TKI's (RAS/Raf, MEK, AKT), mTOR inhibitors and angiogenesis inhibitors (VEGV/VEGFR, PDGF/PDGFR) but bevacizumab will be allowed.
9. Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements to be conducted within 7 days prior to screening:

   * Hemoglobin ≥ 9.0 g/dl
   * Absolute neutrophil count (ANC) ≥ 1,500/mm3
   * Platelet count ≥ 100,000/μl
   * Total bilirubin ≤ 1.5 x upper limit of normal
   * ALT and AST ≤ 2.5 x upper limit of normal (< 5 x upper limit of normal for patients with liver involvement of their cancer)
   * Alkaline phosphatase ≤ 4 x upper limit of normal
   * PT-INR and PTT ≤ 1.5 x upper limit of normal [Patients who are being therapeutically anticoagulated with an agent such as coumadin or heparin will be allowed to participate provided that no prior evidence of underlying abnormality in these parameters exists.]
   * Serum creatinine ≤ 1.5 x upper limit of normal.
10. Signed and dated informed consent before the start of specific protocol procedures.

Exclusion Criteria:

1. History of cardiac disease: congestive heart failure >NYHA class 2; active CAD (MI more than 6 months prior to study entry is allowed); cardiac arrhythmias requiring anti-arrhythmic therapy (beta blockers or digoxin are permitted) or uncontrolled hypertension.
2. Known history of HIV infection or chronic hepatitis B or C
3. Active clinically serious infections (> grade 2 NCI-CTC version 4.02)
4. Prior clinical or radiological evidence of CNS metastases including previously treated, resected, or asymptomatic brain lesions or leptomeningeal involvement by contrast enhanced head CT scan or MRI
5. Patients with seizure disorder requiring medication (such as steroids or anti-epileptics)
6. History of organ allograft
7. Patients with evidence or history of bleeding diathesis
8. Patients undergoing renal dialysis
9. Previous or concurrent cancer that is distinct in primary site or histology from the cancer being evaluated in this study EXCEPT cervical carcinoma in situ, treated basal cell carcinoma, superficial bladder tumours [Ta, Tis & T1] or any cancer curatively treated > 3 years prior to study entry.
10. Pregnant or breast-feeding patients. Women of childbearing potential must have a negative pregnancy test performed within 7 days of the start of treatment. Women enrolled in this trial must use adequate barrier birth control measures during the course of the trial.
11. Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results
12. Any condition that is unstable or could jeopardise the safety of the patient and their compliance in the study
13. Patients unable to swallow oral medications.
14. Patients with intolerance to Paclitaxel.

Excluded therapies and medications, previous and concomitant:

1. Anticancer chemotherapy, hormonotherapy or immunotherapy during the study or within 3 weeks of study entry.
2. Radiotherapy within 3 weeks of start of study drug, palliative radiotherapy will be allowed.
3. Major surgery within 4 weeks of start of study
4. Autologous bone marrow transplant or stem cell rescue within 4 months of study entry
5. Use of biologic response modifiers, such as G-CSF, within 3 week of study entry. [G-CSF and other hematopoietic growth factors may be used in the management of acute toxicity such as febrile neutropenia when clinically indicated or at the discretion of the investigator; however they may not be substituted for a required dose reduction.] [Patients taking chronic erythropoietin are permitted provided no dose adjustment is undertaken within 2 months prior to the study or during the study]
6. Investigational drug therapy outside of this trial during or within 4 weeks of study entry
7. Previous treatment with paclitaxel within 1.line and 2.line palliative therapy (Paclitaxel within (neo-) adjuvant therapy is allowed)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2010-07-01 (Actual); Primary Completion 2014-08-31 (Actual); Study Completion 2014-08-31 (Actual)

PRIMARY OUTCOMES:
Progression free survival (PFS) | app. 3 yrs
  The primary study objective is the proof of efficacy, measured by progression free survival (PFS) in the treatment of metastatic or locally inoperable recurrent breast cancer.
  Progression-free survival (PFS) is defined as the time from randomisation to disease progression or death.

SECONDARY OUTCOMES:
Secondary Efficacy Variables | app. 3 years
  * Clinical benefit (CR+PR+SD)
  * ORR (CR+PR)
  * Time to progression
  * Time to next Treatment (TTT)
  * Overall survival
  * Safety profile

CONTACTS AND LOCATIONS:
Overall Officials: Friedrich Overkamp, Dr. med., Principal Investigator
Locations (1):
- Germany Multiple Sites All Over Germany Recruiting Multiple Sites, Germany Contact: iOMEDICO AG, Freiburg im Breisgau, Germany

REFERENCES:
- [Background] Seidman AD, Berry D, Cirrincione C, Harris L, Muss H, Marcom PK, Gipson G, Burstein H, Lake D, Shapiro CL, Ungaro P, Norton L, Winer E, Hudis C. Randomized phase III trial of weekly compared with every-3-weeks paclitaxel for metastatic breast cancer, with trastuzumab for all HER-2 overexpressors and random assignment to trastuzumab or not in HER-2 nonoverexpressors: final results of Cancer and Leukemia Group B protocol 9840. J Clin Oncol. 2008 Apr 1;26(10):1642-9. doi: 10.1200/JCO.2007.11.6699. PMID 18375893
- [Background] Gradishar W, Kaklamani V, Prasad Sahoo T. A double-blind, randomized, placebo-controlled, Phase 2b study evaluating the efficacy and safety of sorafenib (SOR) in combination with Paclitaxel (PAC) as a first-line therapy in patients with locally recurrent or metastatic breast cancer. Presented at : 32nd Annual San Antonio Breast Cancer Symposium. 2009 Dez 10;(Abstract 44).
- [Derived] Decker T, Overkamp F, Rosel S, Nusch A, Gohler T, Indorf M, Sahlmann J, Trarbach T. A randomized phase II study of paclitaxel alone versus paclitaxel plus sorafenib in second- and third-line treatment of patients with HER2-negative metastatic breast cancer (PASO). BMC Cancer. 2017 Jul 25;17(1):499. doi: 10.1186/s12885-017-3492-1. PMID 28743247